CLINICAL TRIAL: NCT07262398
Title: Effect Of Unilateral Intra-thecal Prilocaine-Fentanyl Versus Bupivacaine-Fentanyl On Post-Operative Spontaneous Voiding Within The Context Of Ambulatory Anesthesia. A Prospective Randomized Double-Blind Controlled Study
Brief Title: Unilateral Intrathecal Bupivacaine Versus Prilocaine on Postoperative Spontaneous Voiding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, professor of anesthesia, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PT (862)
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-08

CONDITIONS: Fast Track Surgery
MeSH Terms: interventions — Prilocaine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: To compare unilateral intrathecal prilocaine versus bupivacaine with added fentanyl in both groups in inguinal hernia repair in the setting of fast-track anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prilocaine (Active Comparator): Prilocaine 40mg (2ml) + fentanyl 25mcg in unilateral spinal anesthesia
  Interventions: Drug: Prilocaine
- Bupivacaine (Active Comparator): Bupivacaine 7.5mg (1.5ml) + fentanyl 25mcg in unilateral spinal anesthesia
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Prilocaine — Prilocaine 40mg (2ml) + fentanyl 25mcg in unilateral spinal anesthesia
  Arms: prilocaine
Drug: Bupivacain — Bupivacaine 7.5mg (1.5ml) + fentanyl 25mcg in unilateral spinal anesthesia
  Arms: Bupivacaine

SUMMARY:
Background: In the context of day-case surgery, the optimal spinal anesthetic should give immediate and effective anesthesia for an appropriate period, followed by rapid regression of sensory and motor blocking, rapid bladder voiding, and little residual effects to allow for early ambulation and discharge. Although bupivacaine is safe and has a low rate of transient neurological symptoms (TNS), the prolonged sensory and motor block is a drawback for use in day-case spinal anesthesia. Similar to lidocaine, prilocaine is a local anesthetic with similar potency and duration of action and has been reported to have a lower incidence of TNS.

Objective: To determine which local anesthetic, Prilocaine with added fentanyl versus bupivacaine with added fentanyl, is better in the setting of fast-track anesthesia in patients undergoing unilateral inguinal hernia.

Material and methods: 70 Patients who were between 18-60 years old male patients, ASA grade I-II, BMI < 35, undergoing elective unilateral inguinal hernia, standard surgical technique (open anterior prosthetic inguinal hernioplasty) inguinal hernia diagnosis is confirmed by ultrasonography, free medical history of micturition disorder, procedure lasting less than 90 minutes, having provided written informed consent signed by the patient or guardian were included. Those patients were divided into two groups. Group Pr (Prilocaine 40mg + fentanyl 25μ) and group Bu (Bupivacaine 7.5mg + fentanyl 25mcg)

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II.
2. BMI < 35 kg/m2.
3. Absence of micturition disorder.
4. Patients scheduled for elective unilateral inguinal hernia with standard surgical technique (open anterior prosthetic inguinal hernioplasty) with previous ultrasonography confirmation of the diagnosis.

Exclusion Criteria:

1. Allergic to any drug being used in the study.
2. ASA III-IV.
3. Suffering from bulky inguinal/inguino-scrotal hernias.
4. Patients with infection at the injection site.
5. Non-cooperative patients.
6. Patients having sensory or motor deficit in lower extremities or history of micturition disorder, abnormal coagulation profile, history of alcohol or substance abuse.
7. contraindications or failure of spinal anesthesia and surgery lasting more than 90 minutes.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — males with no past history of urinary symptoms
Enrollment: 70 (Actual)
Dates: Start 2024-08-03 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
postoperative voiding | first 2 hours postoperatively
  time for the first spontaneous micturition

SECONDARY OUTCOMES:
peak level of spinal anesthesia | 15 minutes
  peak level of spinal anesthesia will be assessed by pinprick after 15 minutes from spinal anesthesia administration to determine the highest dermatome blocked.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data will be provided upon request from the principal investigator
Supporting Information: Study Protocol
Time Frame: 1/12/2025 till 30/12/2026
Access Criteria: researches

REFERENCES:
- [Background] Manish B. Kotwani, Kanchan Rupwate, Prashanth Shivananda, et al. Comparison between high dose hyperbaric Bupivacaine (12.5 mg) alone versus low dose hyperbaric Bupivacaine (7.5mg) with Fentanyl (25 μg) in spinal Anaesthesia for inguinal hernia surgery. Int J Clin Trials. 2016 Aug; 3(3):140-146.
- [Background] Rattenberry W, Hertling A, Erskine R. Spinal anaesthesia for ambulatory surgery. BJA Educ. 2019 Oct;19(10):321-328. doi: 10.1016/j.bjae.2019.06.001. Epub 2019 Aug 13. No abstract available. PMID 33456853